CLINICAL TRIAL: NCT05582811
Title: Riociguat (BAY 63-2521), a Stimulator of Soluble Guanylate Cyclase (sGC) - Cerebral Vasodilation and Headache Induction in Healthy Volunteers
Brief Title: Effect of Riocigaut on Cerebral Vasodilation and Headache Induction in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, MD, Ph.D., DMSc., Chief Consultant Neurologist, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-22020347
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Riociguat 2,5 or 5mg (Experimental): Riociguat dose finding pilot experiment, 2,5mg and 5mg
  Interventions: Drug: Dose Riociguat 2,5 or 5mg
- Riociguat (Active Comparator): Riociguat orally
  Interventions: Drug: Riociguat
- Placebo (Placebo Comparator): Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dose Riociguat 2,5 or 5mg — A selective stimulator of soluble guanylate cyclase (sGC)
  Arms: Dose Riociguat 2,5 or 5mg
Drug: Riociguat — A selective stimulator of soluble guanylate cyclase (sGC)
  Arms: Riociguat
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled cross-over clinical trial aims to investigate the effects of riocigaut on cerebral arteries and headache inducing properties in healthy volunteers.

DETAILED DESCRIPTION:
The investigators believe that activation of sGC could play a role in migraine pathophysiology and propose that stimulation with riociguat causes cranial arterial dilation alongside headache in healthy volunteers.

Twelve healthy volunteers participate at a screening visit, and if eligible, on two separate study days, where participants, in a randomized cross-over fashion, will ingest either riociguat (active comparator arm) or placebo (placebo comparator arm), serving as their own controls. On the two separate study days the investigators will measure change in diameter of superficial temporal artery and middle cerebral artery blood flow velocity and register possible headache until 4 hours after intake of riociguat or placebo. At home participants are expected to fill out a headache diary until 12 hours from intake of riociguat or placebo.

Leading up to the main study described above, the investigators will conduct a pilot dose-finding study (experimental arm) of increasing doses of riociguat, 2,5mg and 5mg respectively, on two separate study days in 5 healthy volunteers, to ensure an appropriate dose is applied in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and receive participant privacy and rights information.
* Male or female participants aged 18-45 years.
* Weight between 50-100kg
* Non-smokers

Exclusion Criteria:

* Any current or previous known primary or secondary headache disorder(s) apart from tension type headache ≤ 1 day per month.
* Headache <48 hours before study start.
* Daily use of any medication except contraceptives. Specifically use of nitrates or nitric oxide donors or phosphodiesterase inhibitors.
* Intake of any pro necessitate medication later than 4 times plasma half-life for the specific drug before study start, except for contraceptives
* Women of child-bearing potential not currently using safe contraceptives. Women of child-bearing potential does not include hysterectomized women and women who have been in menopause for at least 2 years. Safe contraceptives include either IUD, birth control pills, surgical sterilization of the woman, depositary gestagen, barrier prevention or sexual abstinence.
* Pregnant or breastfeeding women
* Positive pregnancy urin screening on screening day or study days.
* A medical history or clinical signs of

  * Hypertension (systolic blood pressure >140mmHg and/or diastolic blood pressure >90mmHg)
  * Hypotension (systolic blood pressure <100mmHg and/or diastolic blood pressure <50mmHg)
* Electrocardiogram (ECG) with any clinically significant abnormalities at screening determined by the investigator, including but not limited to, prolonged PQ or QTc interval, signs of arrythmias, ischemia or left/right ventricle dysfunction/hypertrophy.
* Blood work at screening with signs of anemia.
* Blood work at screening with signs of abnormal kidney and liver function.
* A medical history or clinical signs of cardiovascular disease including cerebrovascular disease.
* A medical history or clinical signs of pulmonary disease.
* A medical history or clinical signs of liver, renal, gastrointestinal, endocrine, hematological or neurological disease.
* A medical history or clinical signs of psychiatric illness or substance abuse
* A medical history or clinical signs of drug or alcohol abuse
* A medical history or clinical signs of disease of any origin that the investigative doctor finds relevant for participation in the study
* A family history of severe cardiac disease.
* Any history of hypersensitivity to riociguat.
* Subjects who do not want information about crucial pathological findings during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in superficial temporal artery (STA) diameter from baseline to 90 minutes in healthy volunteers after receiving riociguat compared to placebo. | 0 - 90 minutes
  Measured by high resolution ultrasonography.

SECONDARY OUTCOMES:
Change in middle cerebral artery (MCA) blood flow velocity in healthy volunteers after receiving riociguat compared to placebo. | 0 - 4 hours
  Measured by transcranial doppler from baseline until 4 hours after intake.
Changes in heart rate in healthy volunteers after receiving riociguat compared to placebo. | 0 - 4 hours
  Measured by heart rate
Incidence of headache (>0 on Numeric Rating Scale (NRS) from 0 to 10, 0="no pain" versus 1-10="pain") in healthy volunteers until 12 hours after receiving riociguat compared to placebo. | 0 - 12 hours
  Data will be collected with a questionnaire.

OTHER OUTCOMES:
Severity of headache, if headache occurs, in healthy volunteers after receiving riociguat compared to placebo, rated on 11-point NRS from 0 ("no pain") to 10 ("worst pain imaginable") from baseline to 12 hours after intake. | 0 - 12 hours
  Data will be collected with a questionnaire.
Headache characteristics, if headache occurs, in healthy volunteers after receiving riociguat compared to placebo, rated from baseline to 12 hours after intake. | 0 - 12 hours
  Data will be collected with a questionnaire.
Reported use of rescue medication if headache occurs, in healthy volunteers, after receiving riociguat compared to placebo. | 0 - 12 hours
  To evaluate need for rescue medication. Data will be collected with a questionnaire.
Time course of STA diameter from baseline until 4 hours after receiving riociguat compared to placebo. | 0 - 4 hours
  Measured by high resolution ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No